CLINICAL TRIAL: NCT01524666
Title: Nutritional Supplementation With Agmatine Sulfate During Small Fiber Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: JFK Medical Center (Other)
Responsible Party: Principal Investigator, Michael Rosenberg, MD, MD, JFK Medical Center
Other Study IDs: AgS-001
Record Dates: First submitted 2012-01-31; First posted 2012-02-02 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Skin Biopsy
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a nonblinded Case-only study that evaluates the effects of Agmatine Sulfate on small fiber peripheral neuropathy. Patients will be started on Agmatine sulfate (a metabolite of Arginine) and monitored for two months. Improvement will be noted on their response to the Neuropathic Pain Questionnaire. Additionally the investigators will note improvement by performing autonomic function testing at the beginning and end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women Ages 18-75 with symptoms of small Fiber Neuropathy and have been diagnosed via autonomic function testing and or skin biopsy

Exclusion Criteria:

* Women who are pregnant or breast feeding, patients with history of substance abuse, and patients with myelopathy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinic patients at JFK Med CTR
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2012-02; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Neuropathic Pain Questionnaire | After 2 months

SECONDARY OUTCOMES:
QSART & ANSAR testing | After 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rosenberg, M.D., Principal Investigator — JFK Medical Center
Locations (1):
- JFK Medical Center, Edison, New Jersey, United States

REFERENCES:
- [Background] Keynan O, Mirovsky Y, Dekel S, Gilad VH, Gilad GM. Safety and Efficacy of Dietary Agmatine Sulfate in Lumbar Disc-associated Radiculopathy. An Open-label, Dose-escalating Study Followed by a Randomized, Double-blind, Placebo-controlled Trial. Pain Med. 2010 Mar;11(3):356-68. doi: 10.1111/j.1526-4637.2010.00808.x. PMID 20447305
- [Derived] Rosenberg ML, Tohidi V, Sherwood K, Gayen S, Medel R, Gilad GM. Evidence for Dietary Agmatine Sulfate Effectiveness in Neuropathies Associated with Painful Small Fiber Neuropathy. A Pilot Open-Label Consecutive Case Series Study. Nutrients. 2020 Feb 23;12(2):576. doi: 10.3390/nu12020576. PMID 32102167